CLINICAL TRIAL: NCT02126345
Title: A Prospective, Observational, Multi-centre, Cohort Study of the MASTER SL Femoral Stem and the DELTA TT Acetabular Cup in Patients With Degenerative Disease of the Hip
Brief Title: MASTER SL Clinical Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-14
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Patients Requiring Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MASTER SL
  Interventions: Device: MASTER SL femoral stem and DELTA TT acetabular cup

INTERVENTIONS:
Device: MASTER SL femoral stem and DELTA TT acetabular cup

SUMMARY:
The purpose of this study is:

* to generate data to evaluate Orthopaedic Data Evaluation Panel (ODEP) rating to support existing short-term clinical results and CE documentation;
* to assess the clinical performance of the MASTER SL femoral stem and the DELTA TT acetabular cup under standard conditions of use;
* to determine any adverse events and assess whether they constitute risks when weighed against the intended performance of the device.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥18 years;
* Radiologically confirmed diagnosis of primary osteoarthritis (OA) of the hip and suitable for primary total hip replacement;
* Life expectancy of >10 years;
* Voluntary written Informed Consent obtained.

Exclusion Criteria:

* Prospect for recovery to independent mobility compromised by known coexistent, medical problems;
* Requiring revision hip replacement;
* Loss of abductor musculature, poor bone stock, or poor skin coverage around the hip joint;
* Previous organ transplant;
* Previous hip replacement (resurfacing or THR) on the contra-lateral side within the last 6 months;
* Previous hip replacement (resurfacing or THR) on the contralateral side and whose outcome is achieving an Oxford Hip score <18 points;
* Body mass index (kg/m2) exceeds 40;
* Active or suspected infection;
* Known sensitivity to device materials;
* Women of childbearing potential who are pregnant, nursing, or planning to become pregnant, and those who do not agree to remain on an acceptable method of birth control throughout the entire study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Requiring Hip Replacement
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Rate of failure | 3 years

SECONDARY OUTCOMES:
Clinical progression measured with HHS score, OHS score, Non-Arthritic Hip Score, EQ-5D-5L | from baseline to all time-points

OTHER OUTCOMES:
Any undesirable side effects | 3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Middleton, MD, Principal Investigator — Royal Bournemouth Hospital NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Royal Bournemouth Hospital NHS Foundation Trust, Bournemouth
  - University Hospital Llandough Cardiff and Vale University Health Board, Cardiff
  - The Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry
  - University Hospital Southampton NHS Foundation Trust, Southampton